CLINICAL TRIAL: NCT04217057
Title: Imaging CCR2 Receptors With 64Cu-DOTA-ECL1i in Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201912003; 1P41EB025815-01 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 64Cu-DOTA-ECL1i-PET/CT (Experimental): -64CU-DOTA-ECL1i-PET/CT imaging consisting of a dynamic scan centered at the level of the known tumor followed by a limited body scan of the head/neck and upper chest will be performed
  Interventions: Drug: 64Cu-DOTA-ECL1i

INTERVENTIONS:
Drug: 64Cu-DOTA-ECL1i — Will be produced by the Cyclotron Facility at Washington University School of Medicine

SUMMARY:
CCR2 is a significant prognostic biomarker in head and neck cancer. Currently there is no clinical biomarker to study CCR2, its prognostic significance or to select patients for CCR2-targeted therapy and to monitor response to such therapy. The investigators have developed a CCR2 specific PET radiotracer based on the peptide, ECL1i (d(LGTFLKC)) and radiolabeled with 64Cu (64Cu-DOTA-ECL1i). The investigators have found that 64Cu-DOTA-ELC1i specific binding has been demonstrated in human head and neck cancer tissue.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years of age or older
* Cytology or biopsy-proven squamous cell head and neck cancer scheduled to be treated with standard of care surgery. Patients who are not surgical candidates should have adequate tissue from tumor biopsy for analysis of CCR2
* Lesion size of at least 1.5 cm (treatment naïve)
* Able to give informed consent
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post menopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 14 hour period immediately prior to administration of 64Cu-DOTA-ECL1i is negative

Exclusion Criteria:

* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 2 years
* Unable to tolerate approximately 90 minutes (total time) of PET/CT imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 64Cu-DOTA-ECL1i-PET/CT
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 64Cu-DOTA-ECL1i-PET/CT
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 62 [56 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 00
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Quality of 64Cu-DOTA-ECL1i-PET/CT Images as Measured by Assessment of Overall Image Quality: 4 Point Scale
Description: -Overall image quality will be graded on a 4 point scale with 1 being the worse and poor quality, not acceptable for diagnostic interpretation and 4 being good image quality, similar to routine clinical studies
Time Frame: At the time of scan (Day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | 64Cu-DOTA-ECL1i-PET/CT
Number analyzed (Participants) | 11
Participants
  Score of 1 | 0
  Score of 2 | 0
  Score of 3 | 0
  Score of 4 | 11

2. Primary Outcome: Diagnostic Quality of 64Cu-DOTA-ECL1i-PET/CT Images as Measured by Presence or Absence of Abnormal 64Cu-DOT-ECL1i Uptake in Pathologically Proven Site of Disease
Time Frame: At the time of scan (Day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | 64Cu-DOTA-ECL1i-PET/CT
Number analyzed (Participants) | 11
Participants
  Presence of abnormal 64Cu-DOT-ECL1i uptake | 11
  Absence of abnormal 64Cu-DOT-ECL1i uptake | 0

3. Primary Outcome: CCR2 Detection Rate of 64Cu-DOTA-ECL1i-PET/CT as Measured by IHC Staining
Description: -Intensity of CCR2 signal in IHC will be assessed by the study pathologist and categorized into 4 categories (0=absent/faint, 1=weak, 2=moderate, 3=strong). Any cells that stained positively with CCR2 will be assessed and the final score will be based on an overall assessment of CCR2 IHC on all of these cells.
Time Frame: At the time of standard of care surgery (estimated to be within 2 weeks of imaging)
Population: One participant did not have tissue avaiable.
Measure: Count of Participants; unit: Participants
Arm/Group | 64Cu-DOTA-ECL1i-PET/CT
Number analyzed (Participants) | 10
Participants
  0=absent/faint | 0
  1=weak | 2
  2=moderate | 5
  3=strong | 3

ADVERSE EVENTS:
Time Frame: Adverse events will be tracked from start of treatment through study discharge (median follow-up of 17 days, full range 7-40 days)
Arm/Group | 64Cu-DOTA-ECL1i-PET/CT
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 64Cu-DOTA-ECL1i-PET/CT (N=11)
Dry mouth (Gastrointestinal disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04217057/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT04217057/ICF_001.pdf